CLINICAL TRIAL: NCT04373018
Title: Comparative Evaluation of Clinical and Radiographic Outcome by Using Three Different Irrigants, Sodium Hypochlorite (NaOCl), Chlorhexidine (CHX) and Combination of CHX+H2O2 in Primary Endodontic Treatment
Brief Title: Evaluation of Three Irrigants, Sodium Hypochlorite, Chlorhexidine and Combination of CHX+H2O2 in Endodontic Treatment.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: anshuyendo
Record Dates: First submitted 2020-04-22; First posted 2020-05-04 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Periapical Periodontitis
Keywords: Sodium hypochlorite; Chlorhexidine; Hydrogen peroxide
MeSH Terms: conditions — Periapical Periodontitis | interventions — Sodium Hypochlorite; Chlorhexidine; Hydrogen Peroxide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sodium hypochlorite (Active Comparator): Procedure/Surgery: Thirty mandibular molars treated with root canal treatment by using Sodium hypochlorite during biomechanical preparation.
  Interventions: Procedure: Sodium hypochlorite
- Chlorhexidine (Active Comparator): Procedure/Surgery: Thirty mandibular molars treated with root canal treatment by using Chlorhexidine during biomechanical preparation.
  Interventions: Procedure: Chlorhexidine
- Chlorhexidine + Hydrogen peroxide (Experimental): Procedure/Surgery: Thirty mandibular molars treated with root canal treatment by using a combination of Chlorhexidine + Hydrogen peroxide during biomechanical preparation.
  Interventions: Procedure: Chlorhexidine + Hydrogen peroxide

INTERVENTIONS:
Procedure: Sodium hypochlorite — Sodium hypochlorite irrigant will be used during biomechanical preparation.
  Arms: Sodium hypochlorite
Procedure: Chlorhexidine — Chlorhexidine irrigant will be used during biomechanical preparation.
  Arms: Chlorhexidine
Procedure: Chlorhexidine + Hydrogen peroxide — Chlorhexidine + Hydrogen peroxide irrigant will be used during biomechanical preparation.
  Arms: Chlorhexidine + Hydrogen peroxide

SUMMARY:
This study will evaluate the synergistic effect of CHX + H2O2 when used as an irrigant during biomechanical preparation.in root canal treatment on periapical healing and compared with Chlorhexidine( CHX) and Sodium Hypochlorite (NaOCl).

DETAILED DESCRIPTION:
After a thorough history, clinical and radiographic examination with all eligibility confirmation, written informed consent will be taken from the patient after explaining the procedure and its associated risks and benefits. Patients randomly allocated to one of the three study groups Sodium hypochlorite (NaOCl), Chlorhexidine (CHX) and combination of (CHX+H2O2). All three irrigants will be used according to standard protocol during biomechanical preparation. Pain analysis will be carried out preoperatively and postoperatively at every 6 hours for 1 day and then every 24 hours till 7 days after the intervention. All the subjects will be followed up for evaluation of clinical and radiographic success at 3, 6 months and 1year.

ELIGIBILITY:
Inclusion Criteria:

* All patients over 18 years of age.
* Mature permanent mandibular molars.
* A radiographic evidence of periapical radiolucency (minimum size > 2mm×2mm) and a diagnosis of pulpal necrosis, as confirmed by the negative response to cold and electrical tests; and absence of bleeding on entering the pulp chamber.

Exclusion Criteria

* Diabetics, immunocompromised patients, pregnant females, any systemic disease.
* Patients with a history of analgesic intake within the past 3 days and antibiotics in the last month.
* Patients with pockets ≥ 4mm or having marginal or furcal bone loss due to periodontitis.
* Non-restorable tooth, fractured, perforated roots and inflammatory root resorption.
* Teeth those are not suitable for rubber dam isolation.
* Primary teeth.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Clinical success | Base line to 1 year.
  Absence of signs and symptoms Absence of tenderness to percussion Tooth mobility of grade 1 or less Absence of associated soft tissue swelling or tenderness to palpation Attachment loss of less than 5mm .
  Two experienced observers with no knowledge of the treatment protocol will independently examine the immediate post obturation and follow up radiographs, mounted side by side, under controlled conditions. The treatment is considered successful only when both clinical and radiographic criteria are met. The worst outcome of an individual root decide the overall outcome for the tooth. In the event of disagreement, the two observers will meet to discuss their findings and came to an agreement.

SECONDARY OUTCOMES:
Radiographic success | Baseline to 1 year
  Absence of periapical alterations (radiolucency at furcal or periapical region) Scoring of each tooth will be done according to the following five point scale (PAI)
  Score Description
  1. Normal Periapical structure
  2. Small changes in bone structure
  3. Changes in bone structure with some mineral loss
  4. Periodontitis with well defined radiolucent area
  5. Severe periodontitis with exacerbating features
Pain assessment | Baseline to 7 days
  Assess the incidence and intensity of pain postoperatively at every 6 hours to 1 day till 7d ays using Visual Analogue scale.Pain intensity will be noted as no pain (0-4mm), mild pain (5-44), moderate pain (45-74mm) and severe pain (75-100mm) on the scale of 0-100mm

CONTACTS AND LOCATIONS:
Overall Officials: Anshu Yadav, Principal Investigator — PGIDS, Rohtak
Locations (1):
- PGIDS, Rohtak, Rohtak, Haryana, India